CLINICAL TRIAL: NCT04822701
Title: A Phase II/III Seamless, Randomized, Double-blind, Placebo-controlled, Parallel-group, Group-sequential Study to Evaluate Efficacy, Safety and Tolerability of BI 767551 for the Treatment of Symptomatic, Non-hospitalized Adults With Mild to Moderate COVID-19.
Brief Title: A Study to Test BI 767551 in People With Mild to Moderate Symptoms of COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: not due to safety reasons
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1487-0001; 2020-005588-29 (EudraCT Number)
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This trial consists of two phases:
  Exploratory Phase II:
  Randomised, double-blind, placebo controlled, doubledummy,Phase II, parallel group design comparing different doses and modes of administration of BI 767551 to placebo.
  Confirmatory Phase III:
  Randomised, double-blind, placebo-controlled, parallel group, Phase III comparing BI 767551 to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase II, Arm 1: Placebo intravenous (i.v.) + placebo inhaled (Placebo Comparator): Single dose of sterile normal saline (NaCl 0.9%) used as placebo for intravenous (i.v.) was administered as intravenous infusion over a period of 60 minutes plus a single inhaled of solvent for dilution of BI 767551 used as placebo for inhalation administered via inhalation through a mouthpiece (Aerogen® Ultra) using a mesh nebulizer (Aerogen® Solo) on Day 1, followed by a 90-day follow-up period. The inhalation procedure was to start approximately 25 min after the start of infusion.
  Interventions: Drug: Placebo intravenous; Drug: Placebo inhaled
- Phase II, Arm 2: BI 767551 10 milligrams (mg)/kilogram (kg) intravenous (i.v.) + placebo inhaled (Experimental)
  Interventions: Drug: BI 767551 intravenous; Drug: Placebo inhaled
- Phase II, Arm 3: BI 767551 40 mg/kg intravenous (i.v.) + placebo inhaled (Experimental)
  Interventions: Drug: BI 767551 intravenous; Drug: Placebo inhaled
- Phase II, Arm 4: Placebo intravenous (i.v.) + BI 767551 250 mg inhaled (Experimental): Single dose of sterile normal saline (NaCl 0.9%) used as placebo for intravenous (i.v.) was administered as intravenous infusion over a period of 60 minutes plus a single inhaled of 250 milligrams (mg) of BI 767551 administered via inhalation through a mouthpiece (Aerogen® Ultra) using a mesh nebulizer (Aerogen® Solo) on Day 1, followed by a 90-day follow-up period. The inhalation procedure was to start approximately 25 min after the start of infusion.
  Interventions: Drug: BI 767551 inhaled; Drug: Placebo intravenous
- Phase III, Arm 1: BI 767551 (medium or high dose infusion) or low dose inhalation (Experimental)
  Interventions: Drug: BI 767551 intravenous
- Phase III, Arm 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo intravenous

INTERVENTIONS:
Drug: BI 767551 intravenous — BI 767551 intravenous
  Arms: Phase II, Arm 2: BI 767551 10 milligrams (mg)/kilogram (kg) intravenous (i.v.) + placebo inhaled; Phase II, Arm 3: BI 767551 40 mg/kg intravenous (i.v.) + placebo inhaled; Phase III, Arm 1: BI 767551 (medium or high dose infusion) or low dose inhalation
Drug: BI 767551 inhaled — BI 767551 inhaled
  Arms: Phase II, Arm 4: Placebo intravenous (i.v.) + BI 767551 250 mg inhaled
Drug: Placebo intravenous — Placebo intravenous
  Arms: Phase II, Arm 1: Placebo intravenous (i.v.) + placebo inhaled; Phase II, Arm 4: Placebo intravenous (i.v.) + BI 767551 250 mg inhaled; Phase III, Arm 2: Placebo
Drug: Placebo inhaled — Placebo inhaled
  Arms: Phase II, Arm 1: Placebo intravenous (i.v.) + placebo inhaled; Phase II, Arm 2: BI 767551 10 milligrams (mg)/kilogram (kg) intravenous (i.v.) + placebo inhaled; Phase II, Arm 3: BI 767551 40 mg/kg intravenous (i.v.) + placebo inhaled

SUMMARY:
This study is open to adults with mild to moderate symptoms of COVID-19 (coronavirus disease). The purpose of this study is to find out whether a medicine called BI 767551 helps people with COVID-19. BI 767551 is an antibody against the coronavirus.

The study has 2 parts.

Part 1 wants to find out the best dose of BI 767551 given as infusion into a vein. It also tests how BI 767551 is taken up by the body when taken via an inhaler. Participants are put into 4 groups by chance. Participants get BI 767551 or placebo once.

* 1 group gets a high dose of BI 767551 as an infusion into a vein
* 1 group gets a low dose of BI 767551 as an infusion into a vein
* 1 group gets BI 767551 via an inhaler
* 1 group gets placebo both as an infusion into a vein and via an inhaler

The placebo infusion and inhaler look like the BI 767551 infusion and inhaler but do not contain any medicine.

Doctors check how BI 767551 reduces the amount of coronavirus. Once the best dose of BI 767551 is found, part 2 of the study tests BI 767551 in a larger group of people. Also, in part 2, the participants get BI 767551 or placebo as an infusion into a vein once. In this part, doctors will check how many people need to be treated in a hospital or die. The results will be compared between the groups.

For each part, participants are in the study for about 13 weeks. During this time, they visit the study site about 8 times and get about 3 remote visits.

The doctors also regularly check participants' health and take note of any unwanted effects of BI 767551.

ELIGIBILITY:
Inclusion criteria phase II and III:

* ≥ 18 years old, males and females
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Documentation of laboratory-confirmed Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, as determined by a molecular test (antigen or nucleic acid) from any respiratory tract specimen (nasopharyngeal (NP) or nasal swab or saliva) collected no more than 72 hours prior to start of treatment
* Patients experienced mild to moderate Coronavirus Disease 2019 (COVID-19)-related symptoms or measured fever for no more than 5 days prior to start of treatment where symptoms are defined by fever, feeling feverish, fatigue, cough, shortness of breath at rest or during activity, sore throat, body pain or muscle pain/ aches, chills, headache, nasal obstruction or congestion, loss of smell or taste, nausea, diarrhea, vomiting, or dysgeusia
* One or more of the following signs/symptoms present on day of start of treatment: fever, feeling feverish, fatigue, cough, shortness of breath at rest or during activity, sore throat, body pain or muscle pain/ aches, chills, headache, nasal obstruction or congestion, loss of smell or taste, nausea, diarrhea, vomiting, or dysgeusia
* Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly

Exclusion criteria phase II and III:

* Body weight of less than 40 kg
* Severe or critical COVID-19 including at least one of

  * Oxygen saturation (SpO2) ≤ 93 % on room air or on their usual level of oxygen supplementation in case of chronic oxygen use
  * Ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) < 300 (in case arterial blood sample was taken)
  * History of hospitalization for COVID-19
  * Current or imminent need for hospitalization or immediate medical attention in the clinical opinion of the site investigator. Does not include patients hospitalized for isolation only
* Receipt of intravenous immunoglobulin within 12 weeks prior to Visit 2
* Receipt of COVID-19 convalescent plasma treatment at any time prior to Visit 2
* Receipt of any SARS-CoV-2 monoclonal antibody treatment at any time prior to Visit 2
* Receipt of SARS-CoV-2 vaccine at any time prior to Visit 2
* Receipt of an investigational product for COVID-19 within 5 half-lives prior to Visit 2
* Receipt of systemic steroids (e.g. prednisone, dexamethasone) within 4 weeks prior to Visit 2 unless used for chronic condition Further exclusion criteria apply.

Exclusion criterion phase III only:

- Previous enrolment in this trial. Patients participating in Phase II are not eligible for Phase III. Re-screening is allowed once, for repeat of Quantitative Reverse Transcription Polymerase chain reaction (RT-qPCR) or antigen SARS-CoV-2 test, if required. The test method used for initial screening (RT-qPCR or antigen) should be used for re-screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Pharmatex Research, Amarillo, Texas
  - Advanced Surgeons and Physicians Network, Houston, Texas
  - Crossroads Clinical Research, Victoria, Texas
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the United States (US) and European Union (EU) for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to evaluate the concept of pharmacological activity of BI 767551 in non-hospitalised patients with mild to moderate COVID-19 symptoms. The study was terminated early. 5 patients total participated in phase II and phase III was not conducted.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo Intravenous (i.v.) + Placebo Inhaled: Single dose of sterile normal saline (NaCl 0.9%) used as placebo was administered as intravenous (i.v.) infusion over a period of 60 minutes plus a single inhaled of solvent for dilution of BI 767551 used as placebo for inhalation administered via inhalation through a mouthpiece (Aerogen® Ultra) using a mesh nebulizer (Aerogen® Solo) on Day 1, followed by a 90-day follow-up period. The inhalation procedure was to start approximately 25 min after the start of infusion.
- Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled: Single dose of sterile normal saline (NaCl 0.9%) used as placebo was administered as intravenous (i.v.) infusion over a period of 60 minutes plus a single inhaled of 250 milligrams (mg) of BI 767551 administered via inhalation through a mouthpiece (Aerogen® Ultra) using a mesh nebulizer (Aerogen® Solo) on Day 1, followed by a 90-day follow-up period. The inhalation procedure was to start approximately 25 min after the start of infusion.
Period: Overall Study
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled
Started | 4 | 1
Treated | 2 | 1
Completed (Completed planned observation time) | 0 | 1
Not Completed | 4 | 0
Not completed — Not treated | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set includes all subjects who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (10.6) | 37.0 (NA) — Only 1 participant was analyzed and no standard deviation can be calculated. | 36.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Log-transformed Nasopharyngeal (NP) swab viral load at baseline [Mean (Standard Deviation); unit: log10 copies / milliliter] — Each viral load result indicates the number of virus copies in a milliliter, and the raw values were log-transformed, resulting in log10 viral load.
  log10 copies / milliliter | 5.24 (2.09) | 7.32 (NA) — Only 1 participants was analyzed and no standard deviation can be calculated. | 5.93 (1.90)

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Time-weighted Change From Baseline in Viral Shedding Over 8 Days in Site Collected Nasopharyngeal (NP) Swabs by Quantitative Reverse Transcription Polymerase Chain Reaction (RT-qPCR)
Description: Time-weighted change from baseline in viral shedding over 8 days in site collected nasopharyngeal (NP) swabs by Quantitative Reverse Transcription Polymerase chain reaction (RT-qPCR), defined as a absolute change from baseline in log10 viral load, is reported.
Time Frame: Up to 8 days
Population: Modified Intention-To-Treat set (mITT): This subject set includes all randomised subjects that received any amount of study drug and who have at least a measurable baseline value (above Lower limit of quantification (LLOQ)) and a second measurement in the first week (up to 7 days after drug intake) of SARS-CoV-2 RNA by site collected nasopharyngeal (NP) swab.
Measure: Mean (Standard Deviation); unit: log10 copies / milliliter
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled
Number analyzed (Participants) | 2 | 1
log10 copies / milliliter | 0.15 (1.25) | -2.84 (NA) — Only 1 participant was analyzed and no standard deviation can be calculated.

2. Secondary Outcome: Phase II: Number of Participants With Loss of Detection of Severe Acute Respiratory Syndrome Coronavirus 2 Ribonucleic Acid (SARS-CoV-2 RNA) by Site Collected NP Swab at Day 4, 8, 15, 22 and 29
Description: Number of participants with loss of detection of Severe acute respiratory syndrome coronavirus 2 ribonucleic acid (SARS-CoV-2 RNA) by site collected NP swab at Day 4, 8, 15, 22 and 29 is report. The "Yes" = loss of detection of SARS-CoV-2 RNA; "No" = SARS-CoV-2 RNA detected; "Missing" = not evaluable.
Time Frame: At Day 4, Day 8, Day 15, Day 22, and Day 29
Population: Treated set (TS): This subject set includes all subjects who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled
Number analyzed (Participants) | 2 | 1
Participants
  Day 4: Yes | 0 | 0
  Day 4: No | 2 | 1
  Day 4: Missing | 0 | 0
  Day 8: Yes | 0 | 0
  Day 8: No | 2 | 1
  Day 8: Missing | 0 | 0
  Day 15: Yes | 1 | 1
  Day 15: No | 1 | 0
  Day 15: Missing | 0 | 0
  Day 22: Yes | 1 | 0
  Day 22: No | 0 | 0
  Day 22: Missing | 1 | 1
  Day 29: Yes | 0 | 0
  Day 29: No | 0 | 0
  Day 29: Missing | 2 | 1

3. Primary Outcome: Phase II: Time-weighted Change From Baseline in Viral Shedding Over 29 Days in Site Collected Nasopharyngeal (NP) Swabs by Quantitative Reverse Transcription Polymerase Chain Reaction (RT-qPCR)
Description: Time-weighted change from baseline in viral shedding over 29 days in site collected nasopharyngeal (NP) swabs by Quantitative Reverse Transcription Polymerase chain reaction (RT-qPCR), defined as a absolute change from baseline in log10 viral load, is reported.
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies / milliliter
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled
Number analyzed (Participants) | 2 | 1
log10 copies / milliliter | -2.09 (1.60) | -4.18 (NA) — Only 1 participant was analyzed and no standard deviation can be calculated.

ADVERSE EVENTS:
Time Frame: From dosing until end of 90-day follow-up period, up to 91 days.
Description: Treated set (TS): This subject set includes all subjects who received any amount of study drug.
Arm/Group | Placebo Intravenous (i.v.) + Placebo Inhaled | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Intravenous (i.v.) + Placebo Inhaled (N=2) | Placebo Intravenous (i.v.) + BI 767551 250 mg Inhaled (N=1)
Parotitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
This trial was prematurely discontinued due to sponsor decision. 4 participants were enrolled in the Phase II "Placebo intravenous (i.v.) + placebo inhaled" group and 1 participant in the "Placebo intravenous (i.v.) + BI 250 mg inhaled" group. No patients were entered in the planned Phase II "BI 10 milligrams (mg)/kilogram (kg) intravenous (i.v.) + placebo inhaled" and "BI 40 mg/kg i.v. + placebo inhaled" groups. Phase III part was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04822701/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT04822701/SAP_001.pdf